CLINICAL TRIAL: NCT04093271
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over, Pilot Study to Investigate the Efficacy of Rest-ZZZ Formula in Healthy Participants With Difficulty Falling Asleep or Staying a Sleep
Brief Title: Investigating the Efficacy of Rest-ZZZ Formula in Healthy Participants With Difficulty Falling Asleep or Staying a Sleep
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LifeSeasons Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 18RSHL
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2019-11

CONDITIONS: Sleep; Healthy
Keywords: Sleep; Healthy; Rest-ZZZ; randomized controlled trial; RCT; dietary supplement; natural health product

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomized to consume Rest-ZZZ, comparator, then placebo (Experimental): Each study product will be consumed as 2 capsules daily for 7 days. Randomized to consume the Rest-ZZZ dietary supplement in Study Period 1, Comparator (Diphenhydramine HCl) in Study Period 2, and Placebo in Study Period 3.
  Interventions: Dietary Supplement: Rest-ZZZ; Drug: Active Comparator - Diphenhydramine HCl; Other: Placebo
- Randomized to consume comparator, placebo, then Rest-ZZZ (Experimental): Each study product will be consumed as 2 capsules daily for 7 days. Randomized to consume the Comparator (Diphenhydramine HCl) in Study Period 1, Placebo in Study Period 2, and the Dietary Supplement, Rest-ZZZ in Study Period 3.
  Interventions: Dietary Supplement: Rest-ZZZ; Drug: Active Comparator - Diphenhydramine HCl; Other: Placebo
- Randomized to consume placebo, Rest-ZZZ, then comparator (Experimental): Each study product will be consumed as 2 capsules daily for 7 days. Randomized to consume Placebo in Study Period 1, Dietary Supplement, Rest-ZZZ in Study Period 2, and Comparator (Diphenhydramine HCl) in Study Period 3.
  Interventions: Dietary Supplement: Rest-ZZZ; Drug: Active Comparator - Diphenhydramine HCl; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Rest-ZZZ — A dietary supplement containing melatonin, valerian root, chamomile, passion flower, GABA, hawthorn berry, and lemon balm
Drug: Active Comparator - Diphenhydramine HCl — DIN 02229960 encapsulated for blinding purposes
Other: Placebo — No active ingredients

SUMMARY:
A randomized, double-blind, placebo-controlled, cross-over pilot study to investigate the efficacy of Rest-ZZZ in healthy participants with difficulty falling asleep or staying a sleep. The study will have 3 study periods. During each study period, eligible participants will consume either Rest-ZZZ, comparator product, or placebo for 7 days during each study period (1 product per study period), with a 1-week washout period in between each period. The primary objective is the comparison in sleep quality using a sleep quality questionnaire from pre-supplement to Day 7 between the Rest-ZZZ, comparator, and placebo. Other study outcomes include the change in quality of life, profile of mood states (POMS), and safety outcomes such as vital signs, clinical chemistry and hematological markers

ELIGIBILITY:
Inclusion Criteria:

1. Has given voluntary, written, informed consent to participate in the study
2. Males and females 25-65 years of age, inclusive
3. BMI of 18-32.5 kg/m2, inclusive
4. Difficulty in falling asleep (taking longer than 30 minutes to fall asleep) or staying asleep, with 2 or more waking episodes in a 7-day period for at least 2 weeks
5. Females participant is not of child bearing potential, defined as females who have had a hysterectomy or bilateral oophorectomy, bilateral tubal ligation, total endometrial ablation or are post-menopausal (natural or surgically with > 1 year since last menstruation) or,

   Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
6. Healthy as determined by laboratory results and medical history and by QI assessment
7. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
8. Agrees to maintain normal diet and exercise routine throughout the study
9. Agrees to maintain current sleep schedule throughout the study
10. Agrees to stay in the current time zone for the duration of the study
11. Agrees to refrain from herbal teas within 2 hours of bedtime, unless currently a part of their night routine for more than 30 days
12. Agrees to refrain from over-the-counter (OTC) products to help with sleep
13. Agrees to refrain from caffeine intake after 3:00 pm during the study
14. Agrees to comply with all study procedures

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
2. Anticipated problems or allergies to any active or inactive ingredients in the investigational products as well as other flowers in the Asteraceae/Compositae family
3. Previous diagnosis of a sleep disorder or use of continuous positive air pressure (C-PAP)
4. Menopausal women with hot flashes
5. Registered with the Canadian National Institute for the Blind (CNIB) and considered as legally blind
6. Currently experiencing vivid nightmares or sleepwalking
7. Have unstable medical conditions such as heart failure, pneumonia, chronic obstructive pulmonary disease (COPD), reflux/gastroesophageal reflux disease (GERD), restless leg syndrome, chronic pain, or disruptive sleep for medical reasons
8. Chronic conditions such as asthma, heartburn, and migraines that consistently interfere with sleep
9. Controlled and uncontrolled hypo- and hypertension
10. Type I and Type II diabetes
11. Current employment that calls for shift work or have worked shift work in the last 3 weeks
12. Travel across 1 or more-time zones in the last 2 weeks and/or is anticipating more travel
13. Clinically significant abnormal laboratory results at screening
14. Use of prescribed medications or any other medications used to help with sleep
15. Use of OTC medications, supplements, food, drinks or products similar to the comparator or Rest-ZZZ to help with sleep. Chamomile, passion flower, valerian root, lemon balm and hawthorn berry ingested as teas and part of daily routine may be included in the study. However, participants will be required to maintain their current routines of consumption until the completion of the study.
16. Evidence or history of clinically significant hematological, renal, endocrine, hepatic, and neurological diseases within the last 5 years as assessed by the QI
17. Autoimmune disease or if immune-compromised (i.e. HIV-positive, use of anti-rejection medication, rheumatoid arthritis, Hepatitis B/C-positive)
18. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow-up that is negative. Volunteers with cancer in full remission for more than 5 years after diagnosis are acceptable after review by QI
19. Diagnosis of any pineal gland abnormalities or have undergone pinealectomy
20. Diagnosis of lower gastrointestinal diseases such as irritable bowel syndrome and inflammatory bowel disease
21. Current or history of bleeding disorders
22. Surgical procedures which may impact the study outcomes within the past 3 months to be assessed by the QI
23. Tobacco use (cigarettes, e-cigarettes, vaporizers, etc.) within 90 days prior to baseline
24. Use of recreational marijuana within 30 days prior to baseline
25. High alcohol intake (average of >2 standard drinks per day or > 10 standard drinks per week)
26. Excessive habitual caffeine consumption (>2 cups coffee or >3 cups caffeinated tea or >2 energy drinks per day) or caffeine intake after 3:00 pm
27. Illicit drug use in the past 6 months as assessed by the QI
28. Participation in clinical trials within 30 days prior to enrollment
29. Blood donation will be assessed on a case-by case basis depending on frequency of donation and hematological and clinical chemistry parameters
30. History of any mental illness that might impair the ability of participants to provide written informed consent
31. Any other condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures, or pose significant risk to the participant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Comparison of change in sleep quality assessed by the sleep quality (SQ) questionnaire between Rest-ZZZ, comparator, and placebo from pre-supplementation to after 7 days of supplementation | 7 days
  The SQ Questionnaire will provide an index for the following parameters: sleep efficiency, perceived sleep debt, and sleep difficulty. In the sleep difficulty section, there are 7 questions asking participants to rate on a scale of 1 to 5 (1 = Strongly Disagree, 2 = Disagree, 3 = No Opinion, 4 = Agree, 5 = Strongly agree). There are 7 questions in the sleep-related quality of life asking participants to rate on a scale of 1 to 5 (1 = Strongly Disagree, 2 = Disagree, 3 = No Opinion, 4 = Agree, 5 = Strongly agree). In both cases, a higher score corresponds to more sleep difficulty and worse sleep-related quality of life (one question in the sleep-related quality of life section has reverse scoring).

SECONDARY OUTCOMES:
Comparison between Rest-ZZZ, comparator, and placebo in the change in quality of life assessed by a quality of life questionnaire from pre-supplementation to after 7 days of supplementation | 7 days
  The quality of life questionnaire will be used to measure discomfort and feelings of well being. This questionnaire has 31 questions assessing different areas in quality of life with various scales.
Comparison between Rest-ZZZ, comparator, and placebo in the change in Profile of Mood States (POMS) questionnaire from pre-supplementation to after 7 of supplementation | 7 days
  The POMS index is used to measure mood states, with its validity well established as its methodology has been used in many clinical trials including other exercise related studies. POMS are a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. Participants will be instructed by a clinic coordinator to respond to the questionnaire based on the past week.

OTHER OUTCOMES:
The incidence of adverse events (AEs) in the Rest-ZZZ, comparator, and placebo groups over the course of the study | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on systolic blood pressure from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on diastolic blood pressure from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on heart rate from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on weight from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on Body Mass Index (BMI) from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on alanine aminotransferase (ALT) levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on aspartate aminotransferase (AST) levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on total bilirubin levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on creatinine levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on sodium levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on potassium levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on chloride levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on hemoglobin levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on hematocrit levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on platelet count levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on mean platelet volume (MPV) levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on red blood cell (RBC) count levels in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on red blood cell (RBC) indices in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on red cell distribution width (RDW) in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on white blood cell (WBC) count in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on neutrophils in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on monocytes in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on eosinophils in the blood from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Rest-ZZZ formula, comparator, or placebo on basophils in the blood from pre-supplementation to Day 7 post-supplementation | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada